CLINICAL TRIAL: NCT06878534
Title: Observational Study Analysing the Transcriptome and Mutational Status of Thyroid Carcinomas of Follicular Origin with Different Degrees of Malignancy
Acronym: TRAMT
Status: Recruiting | Type: Observational
Sponsor: IRCCS SYNLAB SDN (Other)
Collaborators: University Federico II of Naples, Department of Clinical and Surgical Medicine (Unknown)
Responsible Party: Principal Investigator, Marco Salvatore, Prof., IRCCS SYNLAB SDN
Other Study IDs: 3/22
Record Dates: First submitted 2025-03-04; First posted 2025-03-17 (Actual); Last update posted 2025-03-17 (Actual); Status verified 2024-11

CONDITIONS: Thyroid Cancer
Keywords: Thyroid Cancer, miRNA, non coding RNA
MeSH Terms: conditions — Thyroid Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples Without DNA — Plasma, serum and Mononuclear cells from blood samples
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Thyroid cancer patients: Patients with thyroid cancer
- Control subjects: Subjects with non-cancerous thyroid pathology

SUMMARY:
Thyroid cancer (TC) is the most common endocrine malignancy, with well-differentiated thyroid carcinomas (DTCs)-papillary (PTC) and follicular (FTC)-comprising the majority of cases. While DTCs generally have favorable prognoses, a subset progresses to poorly differentiated or anaplastic thyroid carcinoma (ATC), which is highly aggressive. Tumor classification is based on histopathology, invasiveness, and molecular characteristics, with new entities like thyroid tumors of uncertain malignant potential (TT-UMP) and non-invasive follicular thyroid neoplasm with papillary-like nuclear features (NIFTP) refining diagnostic criteria.

Current standard treatments include surgical resection, radioactive iodine therapy, and thyroid hormone replacement. However, some patients develop radioiodine-refractory disease with an increased risk of recurrence and progression. Molecular alterations in the MAPK and PI3K pathways play critical roles in thyroid tumorigenesis, influencing therapeutic response and prognosis. Identifying novel biomarkers for early detection and risk stratification is crucial. Emerging evidence highlights the role of microRNAs (miRNAs) in thyroid cancer progression, functioning as oncogenes or tumor suppressors.

This retrospective case-control study aims to identify novel molecular markers linked to thyroid cancer aggressiveness. Archived formalin-fixed paraffin-embedded (FFPE) tissue and blood samples will be analyzed from patients with varying degrees of PTC and FTC invasiveness. Control samples will be histologically normal thyroid tissue from the same patients.

Next Generation Sequencing (NGS), including RNA-seq and miRNA-seq, will be employed to detect differentially expressed RNA molecules. Validation will be performed using Real-Time PCR in an independent cohort. High-throughput genomic sequencing (Illumina TruSight Oncology 500) will assess mutations, copy number variations, and tumor mutation burden to correlate genetic alterations with malignancy. Variants will be prioritized based on frequency differences in tumor vs. non-tumor populations and functional relevance.

The study will enroll patients with follicular cell-derived thyroid carcinoma. A power analysis indicates that 80 subjects provide >80% statistical power for biomarker identification. Descriptive statistics, parametric/non-parametric tests, and machine learning approaches will analyze transcriptomic and genomic data. Receiver operating characteristic (ROC) curves will assess diagnostic biomarker accuracy, while logistic regression will model associations between molecular alterations and disease severity.

This study aims to uncover molecular mechanisms driving thyroid cancer progression and identify biomarkers for improved risk stratification, early diagnosis, and potential therapeutic targeting. Findings may enhance personalized treatment approaches in thyroid oncology.

ELIGIBILITY:
Inclusion Criteria:

* Patients of either sex aged > 18 years with thyroid cancer of follicular origin.

Exclusion Criteria:

* Patients who do not fit the inclusion criteria.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The study population consists of patients with thyroid carcinoma originating from the follicular thyroid cell at varying degrees of malignancy. For such a retrospective population, considering the study's primary objective of identifying potential tissue biomarkers of pathology, an a posteriori power analysis was performed, considering a paired statistical design of the case-control type, where the control group is afferent to the healthy counterpart of the tissues available in the archives of the same thyroid carcinoma patients.
  For the subgroup analyses associated with the different degrees of invasiveness/aggressiveness, the statistical power associated with the possible clinical stratifications will be assessed before proceeding with the statistical analyses
Sampling Method: Non-Probability Sample
Enrollment: 80 (Estimated)
Dates: Start 2023-03-13 (Actual); Primary Completion 2024-07-30 (Actual); Study Completion 2027-03-31 (Estimated)

PRIMARY OUTCOMES:
Identification of novel molecular biomarkers associated with the progression and aggressiveness of follicular-derived thyroid carcinomas | 1-36 months
  RNA-seq and miRNA-seq on serum samples
Determine genetic alterations hat may contribute to disease progression | 1-36 months
  Identification of mutations, copy number variations, and tumor mutation burden)

SECONDARY OUTCOMES:
Develop of predictive models for improved risk stratification and prognosis | 12-36 months
  Application of machine learning approach to integrate transcriptomic and genomic data

CONTACTS AND LOCATIONS:
Overall Officials: Giovanni Smaldone, Principal Investigator — IRCCS SYNLAB SDN
Locations (1):
- Irccs Synlab Sdn, Naples, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Haugen BR, Alexander EK, Bible KC, Doherty GM, Mandel SJ, Nikiforov YE, Pacini F, Randolph GW, Sawka AM, Schlumberger M, Schuff KG, Sherman SI, Sosa JA, Steward DL, Tuttle RM, Wartofsky L. 2015 American Thyroid Association Management Guidelines for Adult Patients with Thyroid Nodules and Differentiated Thyroid Cancer: The American Thyroid Association Guidelines Task Force on Thyroid Nodules and Differentiated Thyroid Cancer. Thyroid. 2016 Jan;26(1):1-133. doi: 10.1089/thy.2015.0020. PMID 26462967
- [Background] Rossi ED, Locantore P, Bruno C, Dell'Aquila M, Tralongo P, Curatolo M, Revelli L, Raffaelli M, Larocca LM, Pantanowitz L, Pontecorvi A. Molecular Characterization of Thyroid Follicular Lesions in the Era of "Next-Generation" Techniques. Front Endocrinol (Lausanne). 2022 May 12;13:834456. doi: 10.3389/fendo.2022.834456. eCollection 2022. PMID 35634500
- [Background] Xu B, Fuchs T, Dogan S, Landa I, Katabi N, Fagin JA, Tuttle RM, Sherman E, Gill AJ, Ghossein R. Dissecting Anaplastic Thyroid Carcinoma: A Comprehensive Clinical, Histologic, Immunophenotypic, and Molecular Study of 360 Cases. Thyroid. 2020 Oct;30(10):1505-1517. doi: 10.1089/thy.2020.0086. Epub 2020 May 8. PMID 32284020
- [Background] Macerola E, Poma AM, Vignali P, Basolo A, Ugolini C, Torregrossa L, Santini F, Basolo F. Molecular Genetics of Follicular-Derived Thyroid Cancer. Cancers (Basel). 2021 Mar 7;13(5):1139. doi: 10.3390/cancers13051139. PMID 33799953
- [Background] Siegel RL, Miller KD, Fuchs HE, Jemal A. Cancer statistics, 2022. CA Cancer J Clin. 2022 Jan;72(1):7-33. doi: 10.3322/caac.21708. Epub 2022 Jan 12. PMID 35020204